CLINICAL TRIAL: NCT04039269
Title: Could Long Term Memory Created by Preoperative Video Information Reduce Post Operative Behavioral Change?
Brief Title: Long Term Memory Preoperative Preparation Reduce Post Operative Behavioral Change
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Ngamjit Pattaravit, Assistant Professor, Dr, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSUEA2
Record Dates: First submitted 2014-01-08; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Behavior; Agitation
Keywords: Post operative Behavioral Changes; Pediatric; Long term memory; video
MeSH Terms: conditions — Behavior; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Multiple (watch > 3 times) (Active Comparator): Preoperative video information
  Interventions: Other: Preoperative video information
- single (watch 1 time) (Active Comparator): Preoperative video information
  Interventions: Other: Preoperative video information
- conventional (do not watch) (No Intervention): Do not watch video

INTERVENTIONS:
Other: Preoperative video information
  Arms: Multiple (watch > 3 times); single (watch 1 time)

SUMMARY:
The study is designed to test the hypothesis that long term memory created by preoperative video information can reduce the incidence of post operative behavioral changes.

DETAILED DESCRIPTION:
Emergence agitation (EA) and Post operative behavioral change (PHC) are unpleasant experiences occurred in children after general anesthesia (GA). Previous study reported that the patient who had marked EA tended to have new-onset of postoperative maladaptive behavioral changes.Both pharmacologic and non pharmacologic interventions such as preoperative video information, hand held video games were used to reduce preoperative anxiety, EA and Post operative behavioral changes. In term of memory creation, short term memory (STM) was created. Later that the formation of memory trace requires time, and that this trace remains fragile until the long term memory formation process has been completed. In this study, the investigators hypothetize that long term memory created by preoperative video information can reduce the incidence of post operative behavioral changes.

ELIGIBILITY:
Inclusion Criteria:

* outpatient elective surgery
* aged between 3-14 years
* ASA physical status I-II

Exclusion Criteria:

* mental retardation
* patient's telephone contact not available
* emergency case
* having ICU admission plan postoperative

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incidences of post operative behavioral changes | up to3 months post operative period
  Use PHBQ (post operative behavioral questionnaire) Postive for postoperative behavioral change: 10% change from baseline sum score

SECONDARY OUTCOMES:
Incidences of Emergence agitation | evaluate PAED scale in the first 5 minutes after patient arrive PACU
  PAED scale, PAED scale > 10 will be classified as positive for emergence agitation
Parental's anxiety level at induction | Evaluate 15 minutes before start anesthesia induction
  STATE trait anxiety test:
  10% change from baseline sum score will be classify as significant change
Child's anxiety level at induction | mYpas will be evaluated immediately after the patient arrives into the operating room
  mYpas scale: 10% change from baseline sum score will be classify as significant change

CONTACTS AND LOCATIONS:
Overall Officials: Ngamjit Pattaravit, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand